CLINICAL TRIAL: NCT07141056
Title: Impact of Emotional Stress on Immune Checkpoint Inhibitor Treatment Outcomes in Hepatocellular Carcinoma: A Multicohort Clinical Study
Brief Title: The Impact of Emotional Stress on Immunotherapy Outcomes in Liver Cancer Patients: A Multi-Cohort Study
Acronym: SOLACE
Status: Recruiting | Type: Observational
Sponsor: Guilin Medical University, China (Other)
Collaborators: the Affiliated hospital of Guilin medical university, China (Unknown)
Responsible Party: Principal Investigator, Yu Yaqun, Principal Investigator,, Guilin Medical University, China
Other Study IDs: 2024IITLL-51
Record Dates: First submitted 2024-12-22; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: HCC - Hepatocellular Carcinoma; Psychological Distress; Immune Checkpoint Inhibitors (ICIs); Cancer, Treatment-Related; Unresectable Hepatocellular Carcinoma
Keywords: Observational Study; Hepatocellular Carcinoma (HCC); Emotional Distress; Immune Checkpoint Inhibitors; Cancer Immunotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasms, Second Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cohort 1: Unresectable HCC First-line ICI: This group includes participants with unresectable hepatocellular carcinoma who will receive first-line immune checkpoint inhibitor therapy. Participants must have BCLC stage B or C disease and Child-Pugh score A or B (≤7). They will receive standard-of-care immune checkpoint inhibitor therapy according to their physician's choice, either as monotherapy or in combination with other treatments. Emotional distress will be assessed before treatment initiation and during therapy using standardized questionnaires and clinical evaluations. Treatment response will be evaluated every 6-8 weeks using mRECIST criteria.
  Interventions: Other: Psychological Stress Status
- Cohort 2: Resectable HCC Adjuvant ICI: This group includes participants with resectable hepatocellular carcinoma who have undergone curative surgery and will receive adjuvant immune checkpoint inhibitor therapy. They will begin immune checkpoint inhibitor therapy within 4-6 weeks after surgery. Emotional distress will be assessed before starting adjuvant therapy and during treatment. Disease-free survival will be monitored through regular follow-up visits and imaging.
  Interventions: Other: Psychological Stress Status
- Cohort 3: Resectable HCC Neoadjuvant ICI: This group includes participants with resectable hepatocellular carcinoma who will receive immune checkpoint inhibitor therapy before planned surgery. They will receive immune checkpoint inhibitor therapy before surgery, with response assessed using mRECIST criteria. Emotional distress will be evaluated before and during treatment. Pathological complete response will be assessed in surgical specimens.
  Interventions: Other: Psychological stress status

INTERVENTIONS:
Other: Psychological Stress Status — Psychological stress status will be assessed using both self-reported and clinician-rated measures. Participants will be categorized into stressed and non-stressed groups based on the following criteria: Self-reported measures (either): PHQ-9 score ≥ 5 (depression symptoms) and/or; GAD-7 score ≥ 5 (anxiety symptoms) Clinician-rated measures (either): HAMD score ≥ 7 (mild depression) and/or HAMA score ≥ 7 (mild anxiety) Additional assessments: Clinical Global Impression Scale (CGI) EORTC QLQ-C30 (quality of life) Assessment timing: Baseline (before starting immunotherapy) After 2-3 cycles of treatment Every 3 months during follow-up.
  Groups: Cohort 1: Unresectable HCC First-line ICI
Other: Psychological Stress Status — Psychological stress status will be assessed using both self-reported and clinician-rated measures. Participants will be categorized into stressed and non-stressed groups based on the following criteria: Self-reported measures (either): PHQ-9 score ≥ 5 (depression symptoms) and/or; GAD-7 score ≥ 5 (anxiety symptoms) Clinician-rated measures (either): HAMD score ≥ 7 (mild depression) and/or HAMA score ≥ 7 (mild anxiety) Additional assessments: Clinical Global Impression Scale (CGI) EORTC QLQ-C30 (quality of life) Assessment timing: Baseline (before starting immunotherapy) After 2-3 cycles of treatment Every 3 months during follow-up.
  Groups: Cohort 2: Resectable HCC Adjuvant ICI
Other: Psychological stress status — Psychological stress status will be assessed using both self-reported and clinician-rated measures. Participants will be categorized into stressed and non-stressed groups based on the following criteria: Self-reported measures (either): PHQ-9 score ≥ 5 (depression symptoms) and/or; GAD-7 score ≥ 5 (anxiety symptoms) Clinician-rated measures (either): HAMD score ≥ 7 (mild depression) and/or HAMA score ≥ 7 (mild anxiety) Additional assessments: Clinical Global Impression Scale (CGI) EORTC QLQ-C30 (quality of life) Assessment timing: Baseline (before starting immunotherapy) After 2-3 cycles of treatment Every 3 months during follow-up.
  Groups: Cohort 3: Resectable HCC Neoadjuvant ICI

SUMMARY:
The goal of this observational study is to learn if emotional distress affects how well liver cancer treatment works in people receiving immunotherapy. Emotional distress means feeling anxious or depressed. The study aims to answer whether having emotional distress before treatment or changes in emotional distress during treatment affect how well immunotherapy works to treat liver cancer. Researchers will compare participants with and without emotional distress to examine differences in how long the cancer stays under control, treatment response, and overall survival time. Study participants will complete mood and quality of life questionnaires, meet with mental health specialists for emotional assessments, undergo regular blood tests to measure stress hormones, have routine medical check-ups and scans to monitor their cancer status, and be followed for up to 3 years. The study includes three groups of people with liver cancer: those starting immunotherapy for cancer that cannot be removed by surgery, those receiving immunotherapy after surgery, and those receiving immunotherapy before surgery. To be eligible for participation, individuals must be 18 years or older, diagnosed with liver cancer, about to start immunotherapy treatment, and able to complete mood questionnaires.

DETAILED DESCRIPTION:
This multi-center prospective cohort study investigates the relationship between emotional distress (ED) and treatment outcomes in patients receiving immune checkpoint inhibitor (ICI) therapy for hepatocellular carcinoma (liver cancer). Recent research suggests that emotional distress may influence how well cancer treatments work, particularly immunotherapy, but this connection hasn't been well studied in liver cancer patients.

Scientific Background: Liver cancer is a major global health concern, with increasing cases worldwide. While immunotherapy has emerged as a promising treatment option, not all patients respond equally well to this therapy. Understanding factors that might influence treatment success is crucial for improving patient care. Recent studies have shown that emotional distress can affect immune system function, which may impact how well immunotherapy works.

Study Design: The study includes three distinct cohorts of liver cancer patients:

Cohort 1: Patients with unresectable liver cancer starting first-line ICI therapy Cohort 2: Patients receiving ICI therapy after surgery (adjuvant therapy) Cohort 3: Patients receiving ICI therapy before surgery (neoadjuvant therapy)

Comprehensive Assessment Approach:

Emotional distress will be evaluated through multiple methods:

Self-reported questionnaires (PHQ-9 for depression and GAD-7 for anxiety) Professional clinical assessments (Hamilton Depression Scale, Hamilton Anxiety Scale, and Clinical Global Impression Scale) Quality of life measurements Biological markers of stress measured through blood tests

Treatment Monitoring: Participants will receive standard-of-care immunotherapy according to their treating physician's recommendations. The study will not influence treatment decisions but will carefully monitor:

Treatment response through regular imaging Side effects Quality of life Changes in emotional well-being Biological markers of stress and immune function Expected Outcomes and Impact: This study aims to: Determine if emotional distress affects treatment outcomes, Identify which patients might benefit from additional psychological support Understand the biological mechanisms linking stress and treatment response, Develop better strategies for supporting patients during immunotherapy Patient Safety and Support: While this is an observational study that doesn't change standard treatment, we recognize that discussing emotional health can be sensitive. The study includes: Regular monitoring of participants' emotional well-being, Access to mental health professionals if needed, Clear protocols for handling any psychological concerns that arise, Protection of patient privacy and confidentiality Long-term Goals: The findings from this study could lead to: Better ways to identify patients who might need extra support during treatment, New strategies to improve treatment effectiveness, More personalized approaches to cancer care that consider both physical and emotional health, Improved understanding of how psychological factors affect cancer treatment Duration and Follow-up: The study will enroll participants over three years, with each participant followed for up to three years. This allows us to understand both immediate and long-term relationships between emotional well-being and treatment outcomes.

Study Innovation: This is one of the first large-scale studies to: Examine the impact of emotional distress on immunotherapy outcomes in liver cancer, Use both patient self-assessments and professional clinical evaluations, Study this relationship across different stages of treatment.

ELIGIBILITY:
Cohort 1 (SOLACE-1):

Inclusion Criteria:

* Age ≥ 18 years
* Able to complete psychological questionnaires
* Child-Pugh liver function class A
* ECOG performance status ≤ 1
* Signed informed consent
* Expected survival > 3 months
* Diagnosed with unresectable HCC by pathology or imaging
* BCLC stage B or C
* Has at least one measurable lesion (mRECIST)
* About to receive first-line ICI treatment

Exclusion Criteria:

* Currently taking antidepressant or anti-anxiety medications
* Previous diagnosis of psychiatric disorders
* Concurrent malignancy
* Unable to complete psychological assessments
* Previous systemic anti-tumor therapy
* Symptomatic brain metastases
* Child-Pugh score > 7

Cohort 2 (SOLACE-2):

Inclusion Criteria:

* Age ≥ 18 years
* Able to complete psychological questionnaires
* Child-Pugh liver function class A
* ECOG performance status ≤ 1
* Signed informed consent
* Expected survival > 3 months
* Pathologically confirmed HCC after curative surgery
* Pathological stage II or III (AJCC 8th edition)
* Will start adjuvant ICI therapy within 4-6 weeks after surgery
* Expected survival > 12 months

Exclusion Criteria:

* Currently taking antidepressant or anti-anxiety medications
* Previous diagnosis of psychiatric disorders
* Concurrent malignancy
* Unable to complete psychological assessments
* Residual lesions after surgery
* Child-Pugh score B or C

Cohort 3 (SOLACE-3):

Inclusion Criteria:

* Age ≥ 18 years
* Able to complete psychological questionnaires
* Child-Pugh liver function class A
* ECOG performance status ≤ 1
* Signed informed consent
* Expected survival > 3 months
* Diagnosed with resectable HCC by pathology or imaging
* Has at least one measurable lesion (RECIST 1.1)
* About to receive neoadjuvant ICI treatment
* Expected survival > 12 months

Exclusion Criteria:

* Currently taking antidepressant or anti-anxiety medications
* Previous diagnosis of psychiatric disorders
* Severe cardiac, pulmonary, or renal dysfunction
* Concurrent malignancy
* Unable to complete psychological assessments
* Previous systemic anti-tumor therapy
* Symptomatic brain metastases
* Child-Pugh score B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients diagnosed with hepatocellular carcinoma (HCC) who are candidates for immune checkpoint inhibitor therapy. This includes three distinct groups: patients with unresectable HCC who are eligible for first-line immunotherapy (BCLC stage B or C disease), patients with surgically resected HCC who are candidates for adjuvant immunotherapy and patients with potentially resectable HCC who are candidates for neoadjuvant immunotherapy . The study will enroll participants regardless of gender, ethnicity, socioeconomic status, education level, or insurance status. A total of 700 participants will be enrolled across all three cohorts from multiple tertiary hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 24 months
  Time from treatment initiation to disease progression or death
Disease-Free Survival (DFS) | Up to 36 months
  Time from surgery to disease recurrence or death
Pathological Complete Response (pCR) Rate | At time of surgery (approximately 6-8 weeks after neoadjuvant therapy)
  Percentage of participants achieving complete pathological response

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 36 months
  Time from treatment initiation to death from any cause
Objective Response Rate (ORR) | Up to 2 years (assessed every 6-8 weeks from from treatment initiation until disease progression or death from any cause)
  Percentage of participants achieving complete or partial response
Stress Biomarker Levels | From baseline up to 36 months (assessed every 3 months until study completion, disease progression, or death from any cause, whichever occurs first)
  Changes in cortisol and ACTH levels
Safety and Adverse Events | Throughout study duration (up to 36 months)
  Frequency and severity of adverse events
Health-Related Quality of Life measured by EORTC QLQ-C30 Total Score | Baseline, 6 weeks, 9 weeks, then every 12 weeks through study completion (up to 3 years).
  EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-C30) scores. The scale ranges from 0 to 100, where higher scores represent better quality of life for functional scales and global health status, but higher scores represent worse symptoms for symptom scales.
Changes in Depression Scores (PHQ-9) | Baseline, 6 weeks, 9 weeks, then every 12 weeks through study completion (up to 3 years)
  Changes in Patient Health Questionnaire-9 (PHQ-9) depression scores from baseline
Changes in Anxiety Scores (GAD-7) | Baseline, 6 weeks, 9 weeks, then every 12 weeks through study completion (up to 3 years)
  Changes in Generalized Anxiety Disorder-7 (GAD-7) scores from baseline
Changes in Depression Scores (HAMD) | Baseline, 6 weeks, 9 weeks, then every 12 weeks through study completion (up to 3 years)
  Changes in Hamilton Depression Rating Scale (HAMD) scores from baseline
Changes in Anxiety Scores (HAMA) | Baseline, 6 weeks, 9 weeks, then every 12 weeks through study completion (up to 3 years)
  Changes in Hamilton Anxiety Rating Scale (HAMA) scores from baseline

OTHER OUTCOMES:
Association between stress biomarkers and treatment response | Baseline, every 3 months during treatment, and up to 3 years follow-up
  Correlation between stress hormone levels and treatment outcomes

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The Second Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - The Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - The Second Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Shaoyang Central Hospital, Shaoyang, Hunan
  - The First Affiliated Hospital of Shaoyang College, Shaoyang, Hunan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FDA Drug and Device Resources — https://clinicaltrials.gov/fda-links
- See also: MedlinePlus related topics: HCC Stress — https://vsearch.nlm.nih.gov/vivisimo/cgi-bin/query-meta?v%3Aproject=medlineplus&v%3Asources=medlineplus-bundle&query=HCC+STRESS